CLINICAL TRIAL: NCT02800629
Title: Blocking Extracellular Galectin-3 in Patients With Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mark C Fisher, Instructor, HMS, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016P001077
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — citrus pectin

STUDY DESIGN:
Intervention Model Description: Randomized, double blind clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Patients will be given Modified Citrus Pectin twice daily for 12 weeks, and have their change in knee pain as measured by survey instruments assessed
  Interventions: Dietary Supplement: Modified Citrus Pectin
- Control (Placebo Comparator): Patients will be given placebo twice daily for 12 weeks, and have their change in knee pain as measured by survey instruments assessed
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Modified Citrus Pectin — MCP versus placebo
  Arms: Intervention
Dietary Supplement: Placebo
  Arms: Control

SUMMARY:
The proposed study is a pilot, double-blind, randomized clinical trial comparing galectin-3 inhibition with MCP to placebo for the treatment of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Knee pain in at least one knee for more than half the days in the month prior to screening
2. X-rays showing evidence of knee osteoarthritis by Kellgren and Lawrence Score two or three, with definite osteophytes and possible or definite joint space narrowing, consistent with mild to moderate knee osteoarthritis. If both knees are affected, patients would choose the more severe knee for outcomes assessments.
3. Willingness to maintain stable analgesic regimen throughout the study period

Exclusion Criteria:

1. Diagnosis of fibromyalgia
2. Presence of an underlying inflammatory disease in the affected knee, including Rheumatoid Arthritis, Psoriatic Arthritis, Gout, Pseudogout, or other inflammatory disease.
3. Patients who cannot give consent will be excluded, as will patients who cannot speak, read and understand English, as we will not have translated documents, consent forms, and surveys for them.
4. While this supplement is considered very safe and low risk, patients with underlying significant cytopenia (white blood cell count less than 4.0, hemoglobin less than 10, or platelets less than 100), or with impaired renal function (glomerular filtration rate less than 60) or elevated liver enzymes will be excluded as well.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
WOMAC-Knee | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fisher, Principal Investigator — MGH
Locations (1):
- MGH, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No